CLINICAL TRIAL: NCT06490146
Title: Menopause Transition, Sex Hormone Deficiency and Autonomic and Vascular Function
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PT-2024-32769
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Menopause
Keywords: blood pressure; perimenopause; vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: premenopausal women without vasomotor symptoms (VMS)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — this is an observational study

SUMMARY:
This is a longitudinal study to determine the influence of the menopause transition on autonomic and vascular function. PI Keller-Ross has published data demonstrating that postmenopausal females have greater sympathetic neural reactivity during a stressor compared with age-matched males and younger females and males. A paucity of literature exists, however, on the role of the menopause transition in autonomic function because the majority of experimental studies on menopause physiology are cross-sectional and/or focused on older, postmenopausal females .

The influence of age on HTN is robust, whereas the effects of menopause are still unclear. Preliminary data demonstrate a clear association between age and sympathetic activity in females; how the transition through menopause influences these relations, however, remains unknown. The study will enroll 80 midlife (45-55 years of age) females to measure longitudinally the trajectory of autonomic and vascular function during the transition through menopause. The study hypothesizes that through the menopause transition, an increase in sympathetic activity and an impaired baroreflex sensitivity and endothelial function will emerge.

ELIGIBILITY:
Inclusion Criteria:

* Female
* age 45-55 years
* premenopausal
* not using any medications determined to affect autonomic function
* eumenorrheic
* not planning to become pregnant for the duration of participation in the study
* English-speaking, literate, willing and able to provide informed consent.

Exclusion Criteria:

* Diabetes
* pregnant or breastfeeding
* cardiac or pulmonary disorders
* severe obesity (body mass index [BMI] ≥ 40 kg/m 2 )
* hypertension
* obstructive sleep apnea
* current use of heart or blood pressure medications, current use of hormonal contraceptives or other forms of exogenous sex hormones
* report of nicotine/tobacco use in the last six months, report of current alcohol abuse,
* history of treatment with chemotherapy/radiation
* coagulopathy disorders and/or use of anticoagulant medications, and current use of anxiolytics and/or antidepressants.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female, age 45-55 years, premenopausal, not using any medications determined to affect autonomic function, eumenorrheic, not planning to become pregnant for the duration of participation in the study, English-speaking, literate, willing and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2030-08-21 (Estimated); Study Completion 2030-08-21 (Estimated)

PRIMARY OUTCOMES:
MSNA- Burst frequency | up to 12 months
  measured in bursts/min
  Microneurography to measure MSNA: Microneurography is a direct measurement of electrical activity of peripheral sympathetic nerves. A tungsten microelectrode is placed in a peripheral nerve (Figure 8) to record real-time activity from efferent sympathetic vasoconstrictor nerve fibers. MSNA is the gold-standard measure for sympathetic activity
  Participants attend experimental visits annually until they enter perimenopause, at which point they will attend such visits every six months.
MSNA- Burst incidence | up to 12 months
  measured in bursts/100 heartbeats
  Microneurography to measure MSNA: Microneurography is a direct measurement of electrical activity of peripheral sympathetic nerves. A tungsten microelectrode is placed in a peripheral nerve (Figure 8) to record real-time activity from efferent sympathetic vasoconstrictor nerve fibers. MSNA is the gold-standard measure for sympathetic activity
  Participants attend experimental visits annually until they enter perimenopause, at which point they will attend such visits every six months.
MSNA- total activity | up to 12 months
  Microneurography to measure MSNA: Microneurography is a direct measurement of electrical activity of peripheral sympathetic nerves. A tungsten microelectrode is placed in a peripheral nerve (Figure 8) to record real-time activity from efferent sympathetic vasoconstrictor nerve fibers. MSNA is the gold-standard measure for sympathetic activity
  Participants attend experimental visits annually until they enter perimenopause, at which point they will attend such visits every six months.

SECONDARY OUTCOMES:
cardiovagal baroreflex sensitivity: ms/mmHg | up to 12 months
  Cardiovagal baroreflex is estimated by responses in the R-R interval of the ECG to changes in systolic pressure.
  Participants attend experimental visits annually until they enter perimenopause, at which point they will attend such visits every six months.
sympathetic baroreflex sensitivity: bursts/100heartbeats/mmHg | up to 12 months
  Sympathetic baroreflex is estimated by responses in MSNA to changes in diastolic pressure.
  Participants attend experimental visits annually until they enter perimenopause, at which point they will attend such visits every six months.
vascular conductance (mL/100mL tissue/min/mmHg) | up to 12 months
  vascular conductance via venous occlusion plethysmography will be quantified by FBF/mean arterial pressure
  Participants attend experimental visits annually until they enter perimenopause, at which point they will attend such visits every six months.

CONTACTS AND LOCATIONS:
Overall Officials: Manda Keller-Ross, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States